CLINICAL TRIAL: NCT04828005
Title: A Two-part Open Label Study of the Pharmacodynamic Effects of Intranasal Nalmefene Compared to Intranasal Naloxone in Healthy Volunteers Under Steady State Opioid Agonism
Brief Title: Pharmacodynamic Evaluation of Intranasal Nalmefene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opiant Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OPNT003-PD-001
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Pharmacodynamic
MeSH Terms: interventions — nalmefene; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Nalmefene (Experimental): Nalmefene hydrochloride nasal spray, 3mg, 1 spray
  Interventions: Drug: Nalmefene hydrochloride
- Intranasal Naloxone (Active Comparator): Naloxone hydrochloride nasal spray, 4mg, 1 spray
  Interventions: Drug: Naloxone hydrochloride

INTERVENTIONS:
Drug: Nalmefene hydrochloride — 3mg Nasal spray
  Arms: Intranasal Nalmefene
Drug: Naloxone hydrochloride — 4mg Nasal Spray
  Arms: Intranasal Naloxone

SUMMARY:
This study is to determine the pharmacodynamics (the effects of the drug and mechanisms of their action within the body) of Nalmefene when given intranasally (IN; into the nose) compared to intranasal naloxone when given to healthy volunteers under steady state opioid agonism.

DETAILED DESCRIPTION:
Open-label, 2-part study. Part 1 is a pilot study to determine the relationship between opioid agonism and suppression of carbon dioxide induced increases in minute ventilation prior to opioid exposure. Part 2 will be a randomized, 2 period, 2 treatment, crossover study to evaluate the pharmacodynamic effects of intranasal (IN) nalmefene compared to IN naloxone to reverse opioid-induced suppression of carbon dioxide induced increases in minute ventilation, in healthy volunteers with prior opioid exposure.

Both Part 1 and Part 2 of the study will consist of an outpatient Screening Visit taking place 28 days prior to admission, an in-clinic Treatment Phase consisting of a 6 or 7 day inpatient stay, and a Follow-Up Phone Call conducted 3 to 7 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 55 years inclusive
* BMI ranging from 18 to 32 kg/m2, inclusive
* Adequate venous access
* Healthy subjects and non-dependent who are non dependent opioid experienced users, opioid experience defined as exposure to an opioid on at least 1 occasion prior to screening

Exclusion Criteria:

* History of clinically significant disease
* Significant trauma injury, major surgery, open biopsy within 30 days prior to screening
* Subject who has a difficult airway for intubation.
* Following an abnormal diet 4 weeks prior to screening
* Use of over-the-counter medications, dietary supplements, herbal products, vitamins or opioid analgesics 14 days before intervention
* Use of enzyme altering drugs 30 days before intervention
* Use of nasal products 28 days before intervention and throughout the study
* Previous or current opioid, alcohol, or other drug dependence
* Donated or received blood 30 days before intervention
* Women who are pregnant or breastfeeding at screening
* Women of childbearing potential unless surgically sterile or use effective contraception
* Current or recent upper respiratory tract infection
* Allergic to nalmefene or naloxone or known hypersensitivity reaction to plastics.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Searle, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1 Setup and Part 1 Extension Setup were Ventilation Models only; outcome measures were not collected in Part 1. Part 2 participant flow was only reported as one group (i.e., it is not possible to show how many participants received each intervention).
Groups:
- Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone: Subjects received First Treatment (1 Day), followed by Washout (4 Days), followed by Second Treatment (1 Day).
  Treatment in Part 1
  * Healthy volunteers with prior opioid exposure received pretreatment with ondansetron (8 mg, oral) and sodium citrate (30 mL, oral) 30 minutes to 1 hour prior to remifentanil infusion.
  * Subjects started receiving a hypercapnic gas mixture (50% O2, 43% N2, 7% CO2) using a ventilatory response to hypercapnia (VRH) face mask at Time 0 minutes, followed by a remifentanil hydrochloride infusion at Time 5 minutes.
  * Subjects received 4 mg IN naloxone hydrochloride at Time 25 minutes.
  * Remifentanil infusion continued up to Time 115 minutes.
- Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone: Subjects received First Treatment (1 Day) only. Treatment in Part 1 Extension.
  * Healthy volunteers with prior opioid exposure received a naloxone challenge test on the day of clinical admission to ensure the subject was not physically dependent on opioids.
  * Subjects then received pretreatment with famotidine (20 mg IV), ondansetron (8 mg, oral), and sodium citrate (30 mL, oral) 30 minutes to 1 hour prior to remifentanil infusion.
  * Subjects started receiving a hypercapnic gas mixture (50% O2, 43% N2, 7% CO2) using a ventilatory response to hypercapnia (VRH) face mask at Time 0 minutes, followed by a remifentanil hydrochloride infusion at Time 10 minutes.
  * IN naloxone hydrochloride was administered at Time 25 minutes.
  * Remifentanil infusion continued up to Time 146 minutes.
- Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone; Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene: Part 2 was a randomized, 2-treatment crossover study to compare Intranasal Nalmefene to Intranasal Naloxone.
  Subjects received First Treatment (1 Day), followed by Washout (4 Days), followed by Second Treatment (1 Day).
  Treatment in Part 2
  * Healthy volunteers with prior opioid exposure received a naloxone challenge test on the day of clinical admission to ensure the subject was not physically dependent on opioids.
  * After the naloxone challenge test, eligibility review and completion of admission procedures, each subject was randomized to receive either IN nalmefene hydrochloride or IN naloxone hydrochloride in a 2-period crossover manner, with a 4-day washout period between doses.
  * All subjects received pretreatment with famotidine (20 mg IV), ondansetron (8 mg, oral), and sodium citrate (30 mL, oral) 30 minutes to 1 hour prior to remifentanil infusion.
  * All subjects started receiving a hypercapnic gas mixture (50% O2, 43% N2, 7% CO2) using a ventilatory response to hypercapnia (VRH) face mask at Time 0 minutes, followed by a remifentanil hydrochloride infusion at Time 10 minutes.
  * In accordance with the randomization schedule, IN nalmefene hydrochloride (3 mg) or IN naloxone hydrochloride (4 mg) was administered at Time 25 minutes.
  * Remifentanil infusion continued up to Time 146 minutes.
Period: Part 1 Setup: 1st Treatment (1 Day)
Arm/Group | Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone | Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene
Started | 7 | 0 | 0 | 0
Completed | 7 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1 Setup: Washout (4 Days)
Arm/Group | Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone | Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene
Started | 7 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Period: Part 1 Setup: 2nd Treatment (1 Day)
Arm/Group | Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone | Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene
Started | 5 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1 Extension: 1st Treatment (1 Day)
Arm/Group | Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone | Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene
Started | 0 | 8 (In the Part 1 Extension, there was no Washout or 2nd Treatment.) | 0 | 0
Completed | 0 | 8 (In the Part 1 Extension, there was no Washout or 2nd Treatment.) | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2: 1st Treatment (1 Day)
Arm/Group | Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone | Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene
Started | 0 | 0 | 34 | 35
Completed | 0 | 0 | 27 | 32
Not Completed | 0 | 0 | 7 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 1
Not completed — Equipment failure | 0 | 0 | 0 | 1
Period: Part 2: Washout (4 Days)
Arm/Group | Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone | Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene
Started | 0 | 0 | 27 | 32
Completed | 0 | 0 | 25 | 30
Not Completed | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2
Period: Part 2: 2nd Treatment (1 Day)
Arm/Group | Part 1 Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 1 Extension Setup (Ventilation Model): Remifentanil, Then Intranasal Naloxone | Part 2: Intranasal Nalmefene Crossover to Intranasal Naloxone | Part 2: Intranasal Naloxone Crossover to Intranasal Nalmefene
Started | 0 | 0 | 25 | 30
Completed | 0 | 0 | 25 | 27
Not Completed | 0 | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Intranasal Nalmefene: Subjects received First Treatment (1 Day), followed by Washout (4 Days), followed by Second Treatment (1 Day).
  Treatment in Part 1
  * Healthy volunteers with prior opioid exposure received pretreatment with ondansetron (8 mg, oral) and sodium citrate (30 mL, oral) 30 minutes to 1 hour prior to remifentanil infusion.
  * Subjects started receiving a hypercapnic gas mixture (50% O2, 43% N2, 7% CO2) using a ventilatory response to hypercapnia (VRH) face mask at Time 0 minutes, followed by a remifentanil hydrochloride infusion at Time 5 minutes.
  * Subjects received 4 mg IN naloxone hydrochloride at Time 25 minutes.
  * Remifentanil infusion continued up to Time 115 minutes.
- Part 1 Extension: Intranasal Nalmefene: Subjects received First Treatment (1 Day) only. Treatment in Part 1 Extension.
  * Healthy volunteers with prior opioid exposure received a naloxone challenge test on the day of clinical admission to ensure the subject was not physically dependent on opioids.
  * Subjects then received pretreatment with famotidine (20 mg IV), ondansetron (8 mg, oral), and sodium citrate (30 mL, oral) 30 minutes to 1 hour prior to remifentanil infusion.
  * Subjects started receiving a hypercapnic gas mixture (50% O2, 43% N2, 7% CO2) using a ventilatory response to hypercapnia (VRH) face mask at Time 0 minutes, followed by a remifentanil hydrochloride infusion at Time 10 minutes.
  * IN naloxone hydrochloride was administered at Time 25 minutes.
  * Remifentanil infusion continued up to Time 146 minutes.
- Part 2: Intranasal Nalmefene Compared to Intranasal Naloxone: Part 2 was a randomized, 2-treatment crossover study to compare Intranasal Nalmefene to Intranasal Naloxone.
  Subjects received First Treatment (1 Day), followed by Washout (4 Days), followed by Second Treatment (1 Day).
  Treatment in Part 2
  * Healthy volunteers with prior opioid exposure received a naloxone challenge test on the day of clinical admission to ensure the subject was not physically dependent on opioids.
  * After the naloxone challenge test, eligibility review and completion of admission procedures, each subject was randomized to receive either IN nalmefene hydrochloride or IN naloxone hydrochloride in a 2-period crossover manner, with a 4-day washout period between doses.
  * All subjects received pretreatment with famotidine (20 mg IV), ondansetron (8 mg, oral), and sodium citrate (30 mL, oral) 30 minutes to 1 hour prior to remifentanil infusion.
  * All subjects started receiving a hypercapnic gas mixture (50% O2, 43% N2, 7% CO2) using a ventilatory response to hypercapnia (VRH) face mask at Time 0 minutes, followed by a remifentanil hydrochloride infusion at Time 10 minutes.
  * In accordance with the randomization schedule, IN nalmefene hydrochloride (3 mg) or IN naloxone hydrochloride (4 mg) was administered at Time 25 minutes.
  * Remifentanil infusion continued up to Time 146 minutes.
- Total: Total of all reporting groups
Arm/Group | Part 1: Intranasal Nalmefene | Part 1 Extension: Intranasal Nalmefene | Part 2: Intranasal Nalmefene Compared to Intranasal Naloxone | Total
Number analyzed (Participants) | 7 | 8 | 69 | 84
Age, Customized [Mean (Standard Deviation); unit: years] | 28.6 (4.50) | 29.1 (11.05) | 29.1 (7.79) | 29.1 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 21 | 24
  Male | 6 | 6 | 48 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 6 | 57 | 69
  Black or African American | 1 | 2 | 6 | 9
  Asian | 0 | 0 | 2 | 2
  American Indian or Alaskan Native | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Not Reported | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 69 | 84
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.03 (3.338) | 24.48 (3.665) | 25.27 (3.316) | 25.17 (3.317)
Weight [Mean (Standard Deviation); unit: kg] | 79.13 (16.616) | 78.65 (9.735) | 78.30 (14.120) | 78.40 (13.833)
Height [Mean (Standard Deviation); unit: cm] | 178.7 (9.71) | 179.8 (9.38) | 175.6 (10.21) | 176.3 (10.08)

OUTCOME MEASURES:

1. Primary Outcome: Change in Minute Ventilation
Description: Change in minute ventilation from opioid induced nadir
Time Frame: 5 minutes
Measure: Mean (Standard Error); unit: L/min
Groups:
- Intranasal Naloxone: Naloxone hydrochloride nasal spray, 4mg, 1 spray Naloxone hydrochloride: 4mg Nasal Spray
- Intranasal Nalmefene: Nalmefene hydrochloride nasal spray, 3mg, 1 spray Nalmefene hydrochloride: 3mg Nasal spray
Arm/Group | Intranasal Naloxone | Intranasal Nalmefene
Number analyzed (Participants) | 59 | 60
L/min | 3.432 (0.6117) | 5.744 (0.6240)
Statistical Analysis 1: Comparison: Intranasal Naloxone; Test type: Non-Inferiority — Alternative hypothesis: Nalmefene reversal not less than 80% naloxone reversal; p < 0.0009, Mixed Models Analysis

2. Secondary Outcome: Maximum Change in Minute Ventilation
Description: Maximum change in minute ventilation from opioid induced nadir
Time Frame: Up to 2 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
Number analyzed (Participants) | 61 | 60
ng/mL | 6.8 (2.7) | 5.8 (3.0)

3. Secondary Outcome: Time to Maximum Change in Minute Ventilation
Description: Time to maximum change in minute ventilation from opioid induced nadir
Time Frame: Up to 2 hours
Measure: Median (Full Range); unit: hour
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
Number analyzed (Participants) | 61 | 60
hour | 0.50 [0.04 to 2.00] | 0.75 [0.13 to 2.00]

4. Secondary Outcome: Change in Minute Ventilation
Description: Change in minute ventilation from opioid induced nadir
Time Frame: 90 minutes
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
Number analyzed (Participants) | 59 | 56
L/min | 2.71 (0.59) | 2.14 (0.62)

5. Secondary Outcome: Change in Minute Ventilation
Description: Change in minute ventilation from opioid induced nadir
Time Frame: 20 minutes
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
Number analyzed (Participants) | 60 | 59
L/min | 6.79 (0.71) | 5.93 (0.68)

6. Secondary Outcome: Change in Minute Ventilation
Description: Change in minute ventilation from opioid induced nadir
Time Frame: 15 minutes
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
Number analyzed (Participants) | 61 | 59
L/min | 7.12 (0.77) | 5.55 (0.64)

7. Secondary Outcome: Change in Minute Ventilation
Description: Change in minute ventilation from opioid induced nadir
Time Frame: 10 minutes
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
Number analyzed (Participants) | 61 | 59
L/min | 6.58 (0.66) | 4.96 (0.69)

8. Secondary Outcome: Change in Minute Ventilation
Description: Change in minute ventilation from opioid induced nadir
Time Frame: 2.5 minutes
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
Number analyzed (Participants) | 60 | 59
L/min | 2.55 (0.38) | 1.71 (0.53)

ADVERSE EVENTS:
Time Frame: Crossover study adverse event data collected form baseline through to day 6 with a +3 to 7 day follow-up. During the 6 day dosing they took either nalmefene or naloxone on day 1 followed by a 3 day washout and the other dose on day 5
Description: Part 1 Setup and Part 1 Extension Setup were Ventilation Models only; adverse events were not collected in Part 1 for Intranasal Nalmefene nor Intranasal Naloxone. Part 2 is reported.
Arm/Group | Intranasal Nalmefene | Intranasal Naloxone
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 56/61 | 52/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Nalmefene (N=61) | Intranasal Naloxone (N=60)
Nausea (Gastrointestinal disorders) | 24 | 25
Vomiting (Gastrointestinal disorders) | 7 | 14
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 6 | 2
Headache (Nervous system disorders) | 36 | 35
Dizziness (Nervous system disorders) | 11 | 13
Dysgeusia (Nervous system disorders) | 2 | 5
Somnolence (Nervous system disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 10 | 4
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hyperhidosis (Skin and subcutaneous tissue disorders) | 4 | 1
Hot Flush (Vascular disorders) | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT04828005/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT04828005/SAP_001.pdf